CLINICAL TRIAL: NCT03150017
Title: The Impact of an Internet-Delivered Cognitive Behavioural Therapy Pain Management Programme (PMP) on People With Spinal Cord Injuries: A Pilot Study
Brief Title: An Internet-Delivered Pain Management Programme for Spinal Cord Injury Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dearbhla Burke (Other)
Collaborators: Health Informatics Society of Ireland (Unknown); Irish Society of Chartered Physiotherapists (Unknown)
Responsible Party: Sponsor-Investigator, Dearbhla Burke, PhD Candidate, University College Dublin
Organization: University College Dublin (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPIRE2017
Record Dates: First submitted 2017-05-05; First posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Chronic Pain, Widespread; Spinal Cord Injuries
MeSH Terms: conditions — Chronic Pain; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online programme (Experimental): SPIRE The programme consists of six modules over six weeks and is based on cognitive behavioural principles. It comprises psychology sessions using cognitive techniques to identify unhelpful and unrealistic thoughts and beliefs related to pain and to challenge and change them and weekly relaxation audios and a home exercise session. Goal setting by participants is used encouraged throughout the programme to aid the implementation of learned CBT techniques into daily life. Educational sessions are delivered across a range of topics including mechanisms of pain after SCI, explanations of the pain gate control theory and how CBT strategies employed can impact on the perception of pain, discussion of medication use, stress management and pacing strategies for activities of daily living.
  Interventions: Other: SPIRE
- Usual Care (No Intervention): Continue to manage pain using usual care.

INTERVENTIONS:
Other: SPIRE — Online pain management programme.
  Arms: Online programme

SUMMARY:
To establish the effectiveness of an internet-delivered cognitive behavioural therapy pain management programme (CBT-PMP) on people with spinal cord injury pain compared with usual care.

DETAILED DESCRIPTION:
A pilot prospective, single blinded, randomised controlled trial with two arms an internet-delivered CBT-PMP for chronic pain post spinal cord injury (SCI) and usual care.

The CBT-PMP will contain 8 sessions over 8 weeks, with outcomes assessed at baseline, post intervention, and 6 months follow-up.

Participants will be adults with chronic pain (pain > 3 months), regular internet access and not undergoing any other psychological treatments.

Following the study those in the intervention strand will be invited to complete a focus group to explore the subjects' overall experience of the online CBT-PMP.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic or non-traumatic SCI
* Chronic SCI pain of more than three months.
* Discharged from acute hospital and rehabilitation services.
* Males/Females >18years.
* Regular computer and Internet access and working knowledge of the internet.
* Fluency in English (verbal and written).

Exclusion Criteria:

* Those who have completed a PMP before
* Mental health issue which requiring psychiatric management.
* Acute injury, currently under specialist medical care.
* Patients with confounding co-morbidities such as cancer, unstable angina / uncontrolled cardiac arrhythmias/ severe aortic stenosis, acute systemic infection accompanied by fever, systemic/inflammatory diseases eg rheumatoid arthritis/substance abuse/significant mental health issues.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-03-08 (Actual); Primary Completion 2017-08-23 (Estimated); Study Completion 2017-08-23 (Estimated)

PRIMARY OUTCOMES:
Quality of life | Change from baseline to six weeks and three months.
  Quality of life as measured by the WHO QoL Bref

SECONDARY OUTCOMES:
Sleep | Change from baseline to six weeks and three months.
  Sleep quality using the Pittsburgh Sleep Quality Index
Mood | Change from baseline to six weeks and three months.
  Mood measured using the Hospital Anxiety and Depression Scale
Pain | Change from baseline to six weeks and three months.
  Pain measured using the International Spinal Cord Injury Pain Basic Dataset (ISCIPDS:B) (Version 1)
Pain interference | Change from baseline to six weeks and three months.
  Pain interference measured using the brief pain inventory
Pain acceptance | Change from baseline to six weeks and three months.
  Pain acceptance measured using the chronic pain acceptance questionnaire
Patients impression of change | Change from baseline to six weeks and three months.
  Patients impression of change as measured using the Patient's Global Impression of Change

CONTACTS AND LOCATIONS:
Locations (1):
- School of Public Health Physiotherapy and Sports Science, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No